CLINICAL TRIAL: NCT05971550
Title: Clearance of Asymptomatic Pharyngeal Carriage of Neisseria Gonorrhoeae With or Without Ceftriaxone Treatment: Randomized Non-inferiority Study
Acronym: PORTAPHAR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP210080
Record Dates: First submitted 2023-04-14; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-02

CONDITIONS: Neisseria Gonorrhoeae Infection; Asymptomatic Pharyngeal Carriage
MeSH Terms: conditions — Gonorrhea | interventions — Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients : Absence of antibiotic treatment (Experimental)
  Interventions: Other: Absence of antibiotic treatment
- Patients : Ceftriaxone (Active Comparator)
  Interventions: Drug: Ceftriaxone

INTERVENTIONS:
Other: Absence of antibiotic treatment — Absence of antibiotic treatment for at most 3 months after screening for asymptomatic NG pharyngeal infection (treatment if onset of symptoms related to STI or positive PCR at 3 months)
  Arms: Patients : Absence of antibiotic treatment
Drug: Ceftriaxone — Ceftriaxone 1000 mg by parenteral intramuscular route, in a single dose, according to the national recommendations in force, to be repeated if pharyngeal PCR again positive for NG during follow-up
  Arms: Patients : Ceftriaxone

SUMMARY:
Since the use of antibiotics, Neisseria Gonorrhoeae (NG) has acquired progressive resistance to penicillins, sulfonamides, tetracyclines and quinolones. The oropharynx is recognized as an important site for DNA exchange between NG and other commensal Neisseria, allowing NG to acquire new antimicrobial resistance. Despite the worrying data on the emergence of resistant NG, the recommendations remain to systematically treat these infections with ceftriaxone, including asymptomatic pharyngeal localizations. The objective of our study is to evaluate a ceftriaxone sparing strategy in order to limit the emergence of antibiotic resistance.

The primary objective of the study is to evaluate the clearance of Neisseria gonorrhoeae, 3 months after the diagnosis of asymptomatic pharyngeal carriage documented on nucleic acid amplification test (NAAT).

DETAILED DESCRIPTION:
Non-inferiority, multicenter, prospective, randomized open-label study, in two parallel arms, comparing the pharyngeal clearance of Neisseria gonorrhoeae (NG) at 3 months with or without treatment with ceftriaxone.

Experimental group: Absence of antibiotic treatment for at most 3 months after screening for asymptomatic NG pharyngeal infection (treatment if onset of symptoms related to Sexually Transmitted Infection or positive Polymerase chain reaction (PCR) at 3 months)

Control group: Ceftriaxone 1000 mg by parenteral intramuscular route, in a single dose, according to the national recommendations in force, to be repeated if pharyngeal Polymerase chain reaction (PCR) again positive for NG during follow-up.

ELIGIBILITY:
Patients (n=154):

Patient inclusion criteria :

* Adult patient (age ≥ 18 years old)
* Patient consulting for a pharyngeal Neisseria gonorrhoeae Sexually Transmitted Infection (STI) and meeting the following criteria :

  * Positive sample for NAAT by PCR in the pharynx for Neisseria gonorrhoeae dating back a maximum of 7 days (the date of the sample and those of inclusion will be compared) and
  * asymptomatic patient
* Absence of symptoms of other bacterial STIs or other asymptomatic bacterial STIs confirmed on the systematic screening assessment carried out within 7 days before inclusion
* Patient's agreement to use protection or abstinence from all oral sex for 3 months follow-up (experimental group) or for 7 days (control group)
* For men whose female partner(s) are of childbearing age and for women of childbearing age: use of effective contraception (failure rate less than 1% per year) throughout research
* Patient benefiting from a social health security scheme
* Patient having signed a free and informed consent

Patients non-inclusion criteria :

* Minor patient
* Symptomatic patient in the pharynx
* Presence of symptoms of another bacterial STI or of an asymptomatic bacterial STI confirmed on the screening report carried out within 7 days before inclusion
* Antibiotic treatment that may be active on Neisseria gonorrhoeae (C3G, Fluoroquinolones, Macrolides, Cyclins, Aminosides, Penicillins) within 14 days before inclusion
* Hypersensitivity to ceftriaxone, other cephalosporins or to any of the excipients
* History of severe hypersensitivity (e.g. anaphylactic reaction) to another class of antibacterial agents of the beta-lactam family (penicillins, monobactams and carbapenems).
* Contraindication to ceftriaxone
* Contraindication to intramuscular injections
* Person under legal protection, under guardianship or curatorship, person deprived of liberty, under safeguard of justice, subject to psychiatric care, under duress, admitted to a health or social establishment for purposes other than those of research
* Pregnant or breastfeeding woman
* Lack of social health insurance
* Patient included in another interventional study

Partners (n=100) :

Partner Inclusion Criteria :

* Sexual contact of the index case (genito-anal or genito-vaginal, oro-genital or oro-anal or oro-oral relations) in the month preceding the inclusion of the index case
* Adult patient (age ≥ 18 years old)
* Patient benefiting from a social health security scheme
* Patient having signed a free and informed consent

Partner non-inclusion Criteria:

* Minor patient
* Person under legal protection, under guardianship or curatorship, person deprived of liberty, under safeguard of justice, subject to psychiatric care, under duress, admitted to a health or social establishment for purposes other than those of research
* Patient included in another interventional study
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a negative pharyngeal nucleic acid amplification test (NAAT) for Neisseria gonorrhoeae (NG) | 3 months after inclusion

SECONDARY OUTCOMES:
Proportion of patients with a negative pharyngeal nucleic acid amplification test (NAAT) and a negative pharyngeal culture for Neisseria gonorrhoeae (NG) | at 1 month after inclusion
Proportion of patients with negative pharyngeal NG cultures | at 3 months after inclusion
Proportion of patients carrying methicillin-resistant Staphylococcus aureus (MRSA) | at 1 month after inclusion
  Impact of ceftriaxone on the carriage of methicillin-resistant Staphylococcus aureus (MRSA) on the pharyngeal sample
Proportion of patients carrying extended-spectrum beta-lactamase (ESBL)-producing Enterobacteriaceae | at 1 month after inclusion
  Impact of ceftriaxone on the carriage of extended-spectrum beta-lactamase (ESBL)-producing Enterobacteriaceae on the anal sample
Proportion of patients carrying methicillin-resistant Staphylococcus aureus (MRSA) | at 3 months after inclusion
  Impact of ceftriaxone on the carriage of methicillin-resistant Staphylococcus aureus (MRSA) on the pharyngeal sample and extended-spectrum beta-lactamase (ESBL)-producing Enterobacteriaceae on the anal sample
Proportion of patients carrying extended-spectrum beta-lactamase (ESBL)-producing Enterobacteriaceae | at 3 months after inclusion
  Impact of ceftriaxone on the carriage of extended-spectrum beta-lactamase (ESBL)-producing Enterobacteriaceae on the anal sample
Proportion of patients with spontaneous pharyngeal clearance of NG | at 1 month after inclusion
  Analysis of factors associated with spontaneous pharyngeal clearance of NG :
  * Socio-demographic and behavioural characteristics
  * Amount of NG in the pharynx assessed by exploratory semi-quantitative PCR
  * Bactericidal activity of anti-gonococcal antibodies and the production of specific anti-gonococcal antibodies in pharyngeal secretions
Proportion of patients with spontaneous pharyngeal clearance of NG | at 3 months after inclusion
  Analysis of the factors associated with spontaneous pharyngeal clearance of NG :
  * Socio-demographic and behavioural characteristics
  * Amount of NG in the pharynx assessed by exploratory semi-quantitative PCR
  * Bactericidal activity of anti-gonococcal antibodies and the production of specific anti-gonococcal antibodies in pharyngeal secretions
Proportion of partners with NAAT positive for NG | At inclusion of the partner
  Proportion of partners with NAAT positive for NG on at least one of the three sites of infection (pharyngeal, anal, first-void urine or vaginal self-sampling)
Proportion of partners with NG cultures positive | At inclusion of the partner
  Proportion of partners with NG cultures positive on at least one of the three sites of infection (pharyngeal, anal, first-void urine or vaginal self-sampling)
Proportion of partners with NAAT positive for NG | at 1 month after inclusion of the partner
  Proportion of partners with NAAT positive for NG on at least one of the three sites of infection (pharyngeal, anal, first-void urine or vaginal self-sampling)
Proportion of partners with NG cultures positive | at 1 month after inclusion of the partner
  Proportion of partners with NG cultures positive on at least one of the three sites of infection (pharyngeal, anal, first-void urine or vaginal self-sampling)
Proportion of partners with NAAT positive for NG | at 3 months after inclusion of the partner
  Proportion of partners with NAAT positive for NG on at least one of the three sites of infection (pharyngeal, anal, first-void urine or vaginal self-sampling)
Proportion of partners with NG cultures positive | at 3 months after inclusion of the partner
  Proportion of partners with NG cultures positive on at least one of the three sites of infection (pharyngeal, anal, first-void urine or vaginal self-sampling)
Proportion of identical genome between partner and patient | Up to 3 months
Proportion of patients with Resistant NG strains | Up to 3 months
Proportion of partners with Resistant NG strains | Up to 3 months
Proportion of adverse events | Up to 3 months

IPD SHARING:
Plan to Share IPD: Undecided